CLINICAL TRIAL: NCT01556412
Title: Pilot Study of Endoscopic Ultrasound as an Early Diagnostic Tool for Evaluation of Suspected Primary Sclerosing Cholangitis
Brief Title: Endoscopic Ultrasound as an Early Diagnostic Tool for Primary Sclerosing Cholangitis
Status: Completed | Type: Observational
Sponsor: Tischendorf, Jens, M.D. (Individual)
Responsible Party: Sponsor
Other Study IDs: Ti-EUS
Record Dates: First submitted 2012-03-11; First posted 2012-03-16 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Primary Sclerosing Cholangitis
Keywords: endoscopic ultrasound; primary sclerosing cholangitis; EUS; cholestatic hepatopathy
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic hepatopathy suspicious of PSC: All patients with chronic hepatopathy of unknown origin and a high risk of primary sclerosing cholangitis as the underlying disease for chronic hepatopathy.
  This group includes all patients with cholestatic hepatopathy (predominantly elevated gamma-glutamyltransferase and alkalic phosphatase) and positive ANCAs (Anti-neutrophil cytoplasmic antibodies) and/or inflammatory bowel disease in medical history.
  Other explanations of cholestatic hepatopathy (like pancreatic tumor or cholelithiasis) must not be apparent in patients eligible for this study.
  Furthermore, infection oder extrahepatic cholestasis already proven by laboratory results or percutaneous ultrasound, which make endoscopic retrograde cholangiography necessary, are exclusion criteria in this study.

SUMMARY:
Primary sclerosing cholangitis (PSC) is a rare chronic cholestatic liver disease, typically affecting middle aged men and is frequently associated with inflammatory bowel disease. Establishing diagnosis in early stages of cholestatic hepatopathy is still a clinical challenge and based on invasive diagnostic procedures: endoscopic retrograde cholangiography (ERC) or percutaneous liver biopsy are needed when magnetic resonance cholangiopancreaticography remains inconclusive. As these procedures are associated with significant risks for the patient, the goal of this study is to evaluate, if endoscopic ultrasound (EUS) of the biliary tract is a useful diagnostic tool in suspected PSC.

DETAILED DESCRIPTION:
Different parameters of the common bile duct (wall thickness and irregularity, irregularity of the common bile duct and enlarged lymph nodes) are measured in patients with cholestatic hepatopathy of unknown causes via endoscopic ultrasound (EUS).

This EUS of the CBD is performed from the bulbar position in the duodenum and at least 5 cm of bile duct had to be visualized to correctly analyze bile duct structure.

Further diagnostic work-up of these patients is performed following current guidelines, and definite diagnosis is compared with results of EUS parameters measured. Thus, diagnostic yield of EUS in patients with suspected PSC is further evaluated.

ELIGIBILITY:
Inclusion Criteria:

* cholestatic hepatopathy defined by elevation of gamma-GT and alkalic phosphatase and
* elevated pANCA and / or medical history of inflammatory bowel disease

Exclusion Criteria:

* sign of significant intrahepatic cholestasis or any other cause of necessity of cholangiography on transabdominal ultrasound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to a single tertiary clinic center with chronic cholestatic hepatopathy
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2009-03; Primary Completion 2012-05 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Suspicion of PSC in endosonographic ultrasound | From date of endosonographic ultrasound until the date of definite diagnosis of cholestatic hepatopathy, up to 3 months (participants will be followed as outclinic patients in our center for an expected average of 6 weeks until definite diagnosis)
  Endosonographic ultrasound of the common bile duct
  Four different diagnostic parameters evaluated during endosonographic ultrasound are evaluated in predicting primary sclerosing cholangitis:
  * Wall thickening ≥ 1.5 mm
  * Irregular wall structure of the common bile duct
  * Irregular caliber of the common bile duct
  * Lymph nodes proven in the perihilar region of at least 10 mm diameter were defined as enlarged.
  With 2 of 4 criteria positive, patients were classified as suspected diagnostic PSC by means of EUS.

CONTACTS AND LOCATIONS:
Overall Officials: Jens JW Tischendorf, M.D., Principal Investigator — Medical Department III, University Hospital RWTH Aachen
Locations (1):
- Medical Department III, University Hospital RWTH Aachen, Aachen, Northrhine-Westfalia, Germany

REFERENCES:
- [Background] Lutz HH, Tischendorf JJ. Management of primary sclerosing cholangitis. World J Hepatol. 2011 Jun 27;3(6):137-41. doi: 10.4254/wjh.v3.i6.137. PMID 21860672
- [Background] Kirchner GI, Tischendorf JJ, Bleck J, Wagner S, Caselitz M, Klempnauer J, Manns MP, Gebel M. Perihilar lymph nodes in patients with primary sclerosing cholangitis with and without cholangiocellular carcinoma. Scand J Gastroenterol. 2008;43(11):1366-70. doi: 10.1080/00365520802200002. PMID 18609164
- [Background] Mesenas S, Vu C, Doig L, Meenan J. Duodenal EUS to identify thickening of the extrahepatic biliary tree wall in primary sclerosing cholangitis. Gastrointest Endosc. 2006 Mar;63(3):403-8. doi: 10.1016/j.gie.2005.10.040. PMID 16500387